CLINICAL TRIAL: NCT04286399
Title: Asian Diabetes Outcomes Prevention Trial
Acronym: ADOPT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Singapore General Hospital (Other); Mackay Memorial Hospital (Other); National Taiwan University Hospital (Other); Peking University People's Hospital (Other); Medanta, The Medicity, India (Other); Public Health Foundation of India (Other); Putrajaya Hospital, Malaysia (Unknown); Universiti Teknologi Mara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADOPT169609
Record Dates: First submitted 2019-10-16; First posted 2020-02-27 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases | interventions — Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists; Adrenergic beta-Antagonists; Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Treatment Group (Other): High dose of RAASi and beta-blockers (unless contraindicated) as well as preferential use of SGLT2i as per local drug label guidelines on top of standard therapy.
  Interventions: Drug: Renin-angiotensin-aldosterone system inhibitors; Drug: Beta blocker; Drug: SGLT2 Inhibitor - Sodium Glucose Cotransporter Subtype 2 Inhibitor Product
- Control Group (No Intervention): Standard therapy where the use of SGLT2i at randomization is not encouraged but RAASi and beta-blockers (except for maximal dosage) are allowed. Prescription or up-titration of the study drugs listed under Intensive Treatment is not encouraged. If investigators/treating physicians feel that further prescription or up-titration is required, a thorough justification is mandatory. Unless there is clinically irrefutable reason, every attempt should be made to use other blood pressure lowering drugs than RAASi or beta-blockers, as well as glucose lowering drugs than SGLT2i, in the control group.

INTERVENTIONS:
Drug: Renin-angiotensin-aldosterone system inhibitors — Research participants in the intensive therapy arm should be strongly encouraged to follow the intensive treatment strategy. Every attempt should be made to up-titrate RAS-antagonists and beta-blockers (max dosage, unless contraindicated) as well as preferentially use SGLT2i (standard dosage, as required) throughout the trial.
  Other Names: Angiotensin-converting enzyme (ACE) inhibitors; Angiotensin II receptor blockers (ARBs)
  Arms: Intensive Treatment Group
Drug: Beta blocker — Research participants in the intensive therapy arm should be strongly encouraged to follow the intensive treatment strategy. Every attempt should be made to up-titrate RAS-antagonists and beta-blockers (max dosage, unless contraindicated) as well as preferentially use SGLT2i (standard dosage, as required) throughout the trial.
  Arms: Intensive Treatment Group
Drug: SGLT2 Inhibitor - Sodium Glucose Cotransporter Subtype 2 Inhibitor Product — Research participants in the intensive therapy arm should be strongly encouraged to follow the intensive treatment strategy. Every attempt should be made to up-titrate RAS-antagonists and beta-blockers (max dosage, unless contraindicated) as well as preferentially use SGLT2i (standard dosage, as required) throughout the trial.
  Other Names: SGLT2 inhibitors
  Arms: Intensive Treatment Group

SUMMARY:
The aim of this study is to identify patients with DM at high risk of CVD using elevated N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels (>125pg/mL), and (2) intensify therapy using renin-angiotensin system (RAS) antagonists, beta-blockers and sodium glucose co-transporter-2 inhibitors (SGLT2i) for primary prevention of cardiovascular events in this high-risk DM population.

DETAILED DESCRIPTION:
Rationale:

Cardiovascular events are the leading cause of death among patients with diabetes. Early identification of high-risk diabetic (DM) patients for intensification of preventive therapy may prevent cardiovascular events.

Aims:

Among biomarker (N-terminal pro-B-type natriuretic peptide, NT-proBNP)-identified high-risk type 2 DM patients without pre-existing cardiovascular disease, to test if intensive preventive therapy (high dose renin-angiotensin-aldosterone system inhibitors [RAASi], beta-blockade, sodium-glucose co-transporter 2 inhibitors [SGLT2i]) may be associated with reduced cardiovascular events compared to standard of care.

Design:

Prospective multinational randomized open-label, parallel group, active-controlled, two-arm, long-term morbidity and mortality trial involving 5 Asian regions (Singapore, Malaysia, China, Taiwan, India; estimated 6 sites each) with patients followed for 2 years.

Population:

Adults with type 2 DM without known cardiovascular disease (defined as known coronary stenosis > 70%, reduced left ventricular ejection fraction < 40%, or a history of myocardial infarction/coronary revascularization/heart failure hospitalization/stroke/prior non-traumatic lower limb amputation or angioplasty) and with NT-proBNP > 125 pg/mL

Duration:

The goal is to include approximately 2,400 patients. It is estimated that about 3,000 patients with NT-proBNP > 125pg/mL have to be screened. The screen failure rate, for reasons other than NT-proBNP, is anticipated to be approximately 20%. The observation period is planned to last for two years. However, the trial is event driven and will continue until predefined event rate is reached (see sample size calculation). The total trial duration is expected to last for four years (two years of recruitment and a two-year observation period after last patient in). Every patient will remain in the study for two years after randomization.

Visits:

Visit 1:

Pre- Screening

Patients who fulfil the first three pre-screening criteria will proceed for NT-proBNP Point-of-Care (POC) testing:

* Type 2 diabetes for at least 6 months (ADA definition)
* Informed consent
* Check Inclusion/exclusion criteria
* NT-proBNP (assessed through local point of care device) *If the results for NT-proBNP fall > 125pg/mL, the patients will proceed for Full-Screening.

Full- Screening

* Patient enrolment details
* Demographic data
* Patient diary (blood pressure, heart rate, blood glucose) - distribution (optional)
* Vital signs -pulse rate and blood pressure
* Height, weight, waist and hip circumference
* Medical history (DM, cardiovascular, general and behavioural)
* Routine Blood sampling for local laboratory, collected from medical record, if available
* Blood collection for Biomarker analysis (Refer to Section 5.3 and Biospecimen manual)
* Urine sample for Urine Albumin/creatinine ratio, collected from medical record, if available
* Electronic randomization (Section 2.6)
* 12-Lead Electrocardiogram (ECG), collected from medical record, if available (For Singapore sites, ECG values are to be acquired, if not available from medical record)
* EuroQoL questionnaire (EQ-5D-5L)
* Drug prescription assessment
* Health service resource utilisation assessment
* Cardiovascular events assessment
* Baseline Adverse Events assessment
* Echocardiography measurements, collected from medical records, if available (all sites)
* Echocardiography image acquisition (for Singapore and Taiwan sites only - optional)

Interim visits for the treatment group Visit 1-4 is mandatory for all patients, interim visits (between Visits 1-2) only for the intensive treatment group for up-titration of RAASi and beta-blockers and initiation/continuation of SGLT2i. The frequency is up to the treating physician and titration steps. A visit is not mandatory for each titration step.

* Patient diary - collect for assessment and distribute new (optional)
* Vital signs -pulse rate and blood pressure
* Routine blood sampling for local laboratory, collected from medical record, if available
* Drug prescription assessment for further up-titration
* Health service resource utilisation assessment
* Cardiovascular events assessment
* Adverse Events assessment Note: SBP and heart rate should not permanently decrease below 100mmHg and 60bpm respectively.

Visit 2 (3 months ± 1 week)

* Patient diary - collect for assessment and distribute new (optional)
* Vital signs -pulse rate and blood pressure
* Routine Blood sampling for local laboratory, collected from medical record, if available
* Urine sample for Urine Albumin/creatinine ratio, collected from medical record, if available
* 12-Lead Electrocardiogram (ECG), collected from medical record, if available (For Singapore sites, ECG values are to be acquired, if not available from medical record)
* Drug prescription assessment1
* Health service resource utilisation assessment
* Cardiovascular events assessment
* Adverse Events assessment

Visit 3 (12 months ± 2 weeks)

* Patient diary - collect for assessment and distribute new (optional)
* NT-proBNP (assessed through local point of care device)
* Vital signs -pulse rate and blood pressure
* Height, weight, waist and hip circumference
* Routine Blood sampling for local laboratory, collected from medical record, if available
* Blood collection for Biomarker analysis (Refer to Section 5.3 and Biospecimen manual)
* Urine sample for Urine Albumin/creatinine ratio, collected from medical record, if available
* 12-Lead Electrocardiogram (ECG), collected from medical record, if available (For Singapore sites, ECG values are to be acquired, if not available from medical record)
* EuroQoL questionnaire (EQ-5D-5L)
* Drug prescription assessment1
* Health service resource utilisation assessment
* Cardiovascular events assessment
* Adverse Events assessment
* Echocardiography image acquisition (for Taiwan only - optional)

Visit 4: End of Study (24 months ± 2 weeks)

* Patient diary - collect for assessment and distribute new (optional)
* Vital signs -pulse rate and blood pressure
* Height, weight, waist and hip circumference
* Routine Blood sampling for local laboratory, collected from medical record, if available
* Urine sample for Urine Albumin/creatinine ratio, collected from medical record, if available
* 12-Lead Electrocardiogram (ECG), collected from medical record, if available (For Singapore sites, ECG values are to be acquired, if not available from medical record)
* EuroQoL questionnaire (EQ-5D-5L)
* Drug prescription assessment
* Health service resource utilisation assessment
* Cardiovascular events assessment
* Adverse Events assessment

Long-term follow-up (LTFU) (36 and 48 months ± 3 weeks)

* Follow up through telephone contact or population registry (if access allowed) until completion of the study
* Long-term cardiovascular events, mortality and hospitalizations.
* Adverse Events assessment
* For all patients, irrespective of whether they reach these two LTFU time points, a final follow-up should be performed at the end of study

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least six months
* ≥ 40 years of age, men or women
* No known cardiovascular disease ( defined as known coronary stenosis > 70%, reduced left ventricular ejection fraction < 40%, or a history of myocardial infarction/ coronary revascularization/ heart failure hospitalization/ stroke/ prior non-traumatic lower limb amputation or angioplasty)
* NT-proBNP > 125 pg/mL
* Written informed consent

Exclusion Criteria:

* History of hypersensitivity to any of the drugs investigated as well as known or suspected contraindications to the study drugs or previous history of intolerance
* Patients already on a maximum dose of RAASi or beta-blocker
* History of DM ketoacidosis/Type 1 DM
* eGFR < 45ml/min/1.73m2
* Symptomatic hypotension and/or Visit 1 systolic blood pressure (SBP) < 100mmHg.
* Symptomatic bradycardia, high-grade AV blocks (Grade 2 and 3) and/or Visit 1 heart rate (HR) < 60bpm.
* Any disease other than diabetes lowering the patient's life expectancy to less than two years.
* Chronic infections (E.g. chronic cystitis, recurrent urinary tract infections) or malignancies or uncontrolled thyroid disorder or liver disease
* Systemic treatment with corticosteroids.
* Pregnant or nursing women
* Any other clinical condition that might affect patients' safety during trial, at the investigator's discretion.
* Participation in an investigational drug trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2034-06-30 (Estimated)

PRIMARY OUTCOMES:
Combined endpoint based on the first occurrence of cardiovascular death or major adverse cardiovascular event | 48 months
  Stroke/myocardial infarction/heart failures events

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Lam Prof, Study Director — National Heart Centre Singapore
Locations (1):
- Singapore General Hospital (SGH), Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No